CLINICAL TRIAL: NCT00528502
Title: Prevention of Laryngeal Reflexes in Minimal Invasive Parathyroid Surgery by the Use of Topical Lidocaine
Brief Title: Lidocaine Supplement for Minimal Invasive Parathyroid Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to no patient enrollment.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-0147
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Parathyroid Disease
Keywords: Parathyroid Disease; Minimal Invasive Parathyroid Surgery; MIPS; Laryngeal Reflexes; Lidocaine; Saline
MeSH Terms: conditions — Parathyroid Diseases | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Experimental): Saline misted into the air breathe during the surgery.
  Interventions: Drug: Saline
- Lidocaine (Experimental): Lidocaine misted into the air during the surgery.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine is misted into the air that you breathe during the surgery.
  Arms: Lidocaine
Drug: Saline — Saline is misted into the air that you breathe during the surgery.
  Arms: Saline

SUMMARY:
Primary Objective:

1. To determine if the application of lidocaine to the airway will obtund or abolish the laryngeal reflexes. This in turn will lead to a quiescent controlled surgical field.

DETAILED DESCRIPTION:
Lidocaine is a local anesthetic that causes numbness to the throat when misted into the air. This numbness in the throat should stop the urge to clear the throat in the middle of the operation. Therefore, this should stop the interruptions during the surgery.

If you agree to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of 2 groups. Participants in Group 1 will receive the saline mist. This will moisturize and soothe the throat. Participants in Group 2 will receive the lidocaine mist. Lidocaine or saline is misted into the air that you breathe during the surgery. You and your surgeon will not be told which group you were assigned to. At the end of the surgery, your surgeon will answer some questions to help determine if the use of lidocaine or saline is beneficial.

You will be considered off-study once you are sent to the recovery room after surgery.

This is an investigational study. Lidocaine is FDA-approved and commercially available for local anesthesia. If you are in the lidocaine or the saline group. Up to 105 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* All outpatients scheduled for MIPS at the ACB by Dr N Perrier, Dr D Evans and Dr JE Lee.

Exclusion Criteria:

* Patients who are excluded will be any who require elective endotracheal intubation as a preoperative decision by the anesthesia team. These patients will be those with sleep apnea, BMI>35, uncontrolled gastro esophageal reflux.
* Patients who have a history of allergy/hypersensitivity to lidocaine.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Severity of Airway Interruption | Assessment made by surgeon during minimally invasive parathyroidectomy surgery
Quality of Operative Field | Assessment made by surgeon during minimally invasive parathyroidectomy surgery

CONTACTS AND LOCATIONS:
Overall Officials: Spencer Kee, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center official web site — http://www.mdanderson.org